CLINICAL TRIAL: NCT01307618
Title: A Randomized Phase II Study of Multipeptide Vaccination With or Without IL-12, Then Combined With Regulatory T Cell Depletion Using Daclizumab in Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy With or Without Recombinant Interleukin-12 Followed by Daclizumab in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of clinical efficacy and lack of drug supply, trial was closed early and correlative studies were not pursued further.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02580; NCI-2011-02580 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-10-324-B; CDR0000696233; 10-324-B (Other: University of Chicago Comprehensive Cancer Center); 8445 (Other: CTEP); P30CA014599 (NIH); N01CM00071 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — MAGEA3 protein, human; Interleukin-12 Subunit p35; MART-1 Antigen

ARMS (2):
- Arm I (vaccine therapy) (Experimental): Patients receive vaccination comprising recombinant MAGE-3.1 antigen, MART-1 antigen, gp100 antigen, and NA17-A2 peptide emulsified with Montanide ISA-51 ID or SC on days 1, 22, and 50.
  Interventions: Biological: NA17.A2 Peptide Vaccine; Biological: Recombinant MAGE-3.1 Antigen; Biological: MART-1 Antigen; Other: Laboratory Biomarker Analysis
- Arm II (vaccine therapy, IL-12) (Experimental): Patients receive vaccination as in arm I with an admixture of IL-12 ID or SC on days 1, 22, and 50.
  Interventions: Biological: NA17.A2 Peptide Vaccine; Biological: Recombinant MAGE-3.1 Antigen; Biological: Recombinant Interleukin-12; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: NA17.A2 Peptide Vaccine — Given SC or ID
  Other Names: NA17.A2
Biological: Recombinant MAGE-3.1 Antigen — Given SC or ID
  Other Names: MAGE-3; MAGE-3.1
Biological: Recombinant Interleukin-12 — Given SC or ID
  Arms: Arm II (vaccine therapy, IL-12)
Biological: MART-1 Antigen — Given SC or ID
  Other Names: Antigen LB39-AA; Antigen SK29-AA; MART-1 Tumor Antigen
  Arms: Arm I (vaccine therapy)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well giving vaccine therapy together with or without recombinant interleukin-12 followed by daclizumab works in treating patients with melanoma that has spread to other places in the body. Vaccines made from peptides or antigens may help the body build an effective immune response to kill tumor cells. Recombinant interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating white blood cells to kill melanoma cells. Monoclonal antibodies, such as daclizumab, may decrease the number of regulatory T cells (T cells that suppress the activation of the immmune system) and may lead to a better immune response against melanoma. It is not yet known whether vaccine therapy is more effective with interleukin-12 and daclizumab in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if admixture of IL-12 (recombinant interleukin-12) with vaccine emulsion will increase the frequency of vaccine-induced cluster of differentiation (CD)8+ T cells in the blood.

II. To determine if administration of daclizumab will deplete CD4+CD25+ regulatory T cells from the peripheral and potentiate specific immune responses induced by vaccination.

III. To determine if vaccination +/- daclizumab will be safe in this patient population.

SECONDARY OBJECTIVES:

I. To determine if vaccination +/- daclizumab will have clinical activity in patients with advanced melanoma.

II. To determine if clinical response may be associated with particular gene expression profiles in the tumor microenvironment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive multipeptide vaccination comprising recombinant MAGE-3.1 antigen, MART-1 antigen, gp100 antigen, and NA17-A2 peptide emulsified with Montanide ISA-51 intradermically (ID) or subcutaneously (SC) on days 1, 22, and 50.

ARM II: Patients receive vaccination as in arm I with an admixture of recombinant interleukin-12 (IL-12) on days 1, 22, and 50.

In both arms, patients are evaluated for immune response. Patients with partial response or stable disease may be immunized for up to a maximum of 1 year. Patients with complete response may be treated with 1 additional course of 3 vaccinations.

EXPANDED COHORT: Additional patients are accrued to the arm with higher immune response and receive daclizumab IV over 15 minutes on day -7. Patients then receive vaccination as in arm I or arm II on days 1, 22, and 50 in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 8 weeks until disease progression and then at least every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed melanoma with evidence of metastatic disease either by radiologic or physical examination

  * In-transit metastases are allowed
  * Biopsy should be performed to reconfirm the diagnosis in cases of doubt
* Patients must have measurable disease

  * For computed tomography (CT) imaging, this is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
  * For cutaneous lesions, these must be measurable with a ruler and documented photographically with a ruler in place
* There are no limits on the number of prior therapies; patients must not have received a vaccine containing any of the melanoma antigen peptides, nor previously received daclizumab; at least 4 weeks must have passed since prior chemotherapy or radiation therapy (6 weeks for BCNU [carmustine] or mitomycin C)
* Life expectancy greater than or equal to 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky ≥ 80%)
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100,000/mcL
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) ≤ 2 x institutional ULN
* Lactate dehydrogenase (LDH) < 1.25 x ULN
* Human leukocyte antigen (HLA) typing: patient must express HLA-A2, either by flow cytometry or by standard HLA typing
* Patient must agree to undergo biopsy of accessible tumor before and after therapy, when feasible, to study tumor cell properties and characteristics of immune cells; if a biopsy cannot be done, then a prior pathologic specimen from the patient must show tumor cells that are positive for melanosome specific antigen (HMB45) and MLANA (MelanA); the tumor must express at least 2 antigens in the vaccine for the patient to be eligible
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, or abstinence) prior to study entry, for the duration of treatment, and for 2 months after completion of treatment; a pregnancy test must be done and be negative for women of child-bearing potential; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, biological or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Presence of untreated brain metastases; all patients must undergo brain imaging as part of the pre-study evaluation; only patients with no brain metastases, or with brain lesions successfully treated by stereotactic radiation or surgical removal without progression at 28-day follow-up and off corticosteroids for 4 weeks, will be eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition IL-12 or other agents used in the study
* Concurrent systemic corticosteroids (except physiologic replacement doses) or other immunosuppressive drugs (eg. cyclosporin A)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with IL-12; women of child-bearing age must be tested for urinary or serum beta-human chorionic gonadotropin (HCG)
* Patients with intrinsic immunosuppression, including seropositivity for human immunodeficiency virus (HIV) antibody; patients should be tested for HIV; HIV-positive patients are ineligible
* Psychiatric illness that may make compliance to the clinical protocol unmanageable or may compromise the ability of the patient to give informed consent; patients with clinical evidence of dementia should have a competent designee participate in decision making
* Serious concurrent infection, including active tuberculosis, hepatitis B, or hepatitis C; patients should be tested for hepatitis B surface antigen and hepatitis C antibody; patients who are hepatitis C antibody (Ab) positive can be eligible if they are polymerase chain reaction (PCR)-negative
* Active or history of autoimmune disease including but not limited to: rheumatoid arthritis (rheumatoid factor [RF]-positive with current or recent flare), inflammatory bowel disease, systemic lupus erythematosis (clinical evidence with antinuclear antibody [ANA] 1:80 or greater), ankylosing spondylitis, scleroderma, multiple sclerosis, autoimmune hemolytic anemia, and immune thrombocytopenic purpura; seropositivity alone will not be considered active autoimmunity; patients with immune-mediated hypothyrodisim and/or vitiligo are allowed
* Active gastrointestinal bleeding or uncontrolled peptic ulcer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajewski, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.86 (12.55) | 66.16 (15.11) | 62.01 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Vaccine-induced CD8+ T Cells Assessed by Enzyme-linked Immunospot (ELISPOT)
Description: Data before treatment and after 3 vaccines will be assessed using paired t-tests within each cohort as well as a two-sample t-test of the mean post-treatment levels between cohorts. Repeated measures analysis of variance or mixed effects models will be utilized to further characterize changes in the levels of circulating T cells over time.
Time Frame: Up to 4 years
Population: Due to lack of clinical efficacy and lack of drug supply, trial was closed early and frequency of vaccine-induced CD8+T cells was not measured.
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Absolute Number of CD4+CD25+FoxP3+ Regulatory T Cells From Peripheral Blood
Description: Descriptive statistics and paired t-tests will be generated to describe the frequency and absolute number of CD4+CD25+FoxP3+ cells before and after daclizumab, and also at subsequent time points. Repeated measures of analysis of variance and mixed effects models will be used to further evaluate change in numbers over time, and to compare these changes between cohorts.
Time Frame: Up to 4 years
Population: Due to lack of clinical efficacy and lack of drug supply, trial was closed early and absolute number of CD4+CD25+FoxP3+Regulatory T Cells from peripheral blood was not measured.
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Type and Grade of Toxicity Incidents Assessed by Common Toxicity Criteria Version 4.0 (CTCAE v4.0)
Time Frame: Up to 4 years
Population: Patients who experienced any adverse event were counted.
Measure: Number; unit: participants
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 5 | 5
participants
  Abdominal pain (Grade 1) | 1 | 0
  Anxiety (Grade 1) | 1 | 1
  Chills (Grade 1) | 1 | 0
  Cough (Grade 1) | 1 | 1
  Diarrhea (Grade 1) | 1 | 0
  Dyspnea (Grade 1) | 1 | 0
  Erythema multiforme (Grade 1) | 1 | 0
  Fatigue (Grade 1) | 3 | 2
  Infections (Grade 1) | 1 | 0
  Injection site reaction (Grade 1) | 4 | 2
  Pruritus (Grade 1) | 1 | 0
  Rectal hemorrhage (Grade1 ) | 1 | 0
  Rectal pain (Grade 1) | 1 | 0
  Arthralgia (Grade 1) | 0 | 1
  Bone pain (Grade 1) | 0 | 1
  Death NOS (Grade 5) | 0 | 1
  Dehydration (Grade 1) | 0 | 1
  Dyspnea (Grade 2) | 0 | 1
  Headache (Grade 1) | 0 | 1
  Hypoalbuminemia (Grade 1) | 0 | 1
  Hypophosphatemia (Grade 1) | 0 | 1
  Pain (Grade 1) | 0 | 1
  Pleuritic pain (Grade 1) | 0 | 1
  Proteinuria (Grade 1) | 0 | 1
  Psychiatric disorders (Grade 2) | 0 | 1

4. Secondary Outcome: Progression-free Survival Assessed by Modified World Health Organization (WHO) Criteria
Description: Median progression-free survival and the associated 95% confidence limits will be derived using the procedure described in Brookmeyer and Crowley.
  The criteria for progressive disease are 1) appearance of new lesions, 2) 25% increase in the sum of the product of the largest perpendicular diameters of the indicator lesions, or 3) reappearance of any tumor.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 5 | 5
days | 130 [77 to NA] — The upper limit of the 95% confidence interval was not reached. | 64 [63 to NA] — The upper limit of the 95% confidence interval was not reached.

5. Secondary Outcome: Overall Survival Assessed by Modified WHO Criteria
Description: Median overall survival and the associated 95% confidence limits will be derived using the procedure described in Brookmeyer and Crowley.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 5 | 5
days | 804 [NA to NA] — The 95% confidence interval was not reached. Only one patient died and others were censored. | 199 [92 to NA] — The upper limit of 95% confidence interval was not reached.

6. Secondary Outcome: Gene Expression Profiles
Description: Gene cluster analysis will be performed using deoxyribonucleic acid (DNA)-Chip Analyzer (dCHIP) software and comparisons will be made before and after treatment in each individual patient, and between responders and non-responders. Attempts will be made to identify gene expression profiles that correlate with clinical outcome.
Time Frame: Up to 4 years
Population: Due to lack of clinical efficacy and lack of drug supply, trial was closed early and gene expression profiles was not measured.
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Vaccine Therapy) | Arm II (Vaccine Therapy, IL-12)
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Vaccine Therapy) (N=5) | Arm II (Vaccine Therapy, IL-12) (N=5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Vaccine Therapy) (N=5) | Arm II (Vaccine Therapy, IL-12) (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 3 | 3
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Injection site reaction (General disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less